CLINICAL TRIAL: NCT00517140
Title: Vaginal Birth After Caesarean Section - Effect on Maternal Psychosocial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2003.118; HARECCTR0500014
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Pregnancy; Cesarean Section; Uterine Rupture
Keywords: Pregnancy women with a scarred uterus due to previous caesarean section
MeSH Terms: conditions — Uterine Rupture

INTERVENTIONS:
Procedure: Repeat Caesaen section
Procedure: vaginal delivery

SUMMARY:
The incidence of caesarean section has reached 15-20% in most developed countries. Encouraging vaginal birth after caesareans section (VBAC) has been considered a key component of a strategy to reduce the caesarean section rate. Most medical literature has focused on the efficacy of VBAC in reducing the caesarean section rate and the physical safety of successful VBAC. However, 30%-40% of these women fail to achieve a vaginal delivery. Little is known about how the uncertainty of labour outcome and a failed VBAC impact on the psychosocial function of these women. We propose to study a cohort of women with a prior caesarean section and presenting with a subsequent pregnancy for care. After consent and recruitment, these subjects will be randomly assigned to have a repeat caesarean section or VBAC. The medical outcomes, overall satisfaction of the subjects with the care they received, and the short-term psychosocial function of these subjects will be studied. The result of this study will provide important information that would be useful in assisting women to decide the mode of delivery after a prior caesarean section.

ELIGIBILITY:
Inclusion Criteria:

All women who:

* Have one prior caesarean section
* No prior vaginal delivery and
* Agree for either vaginal delivery or elective caesarean section

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2003-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
pscyiatric morbidity | after delivery

SECONDARY OUTCOMES:
Psychosocial function | 3 and 6 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tze Kin Lau, Prof, Principal Investigator — Department of Obstetrics and Gynaecology, The Chinese Univerisity of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Prince of Wales Hospital, Hong Kong, China